CLINICAL TRIAL: NCT04215523
Title: Replication of the Dapagliflozin Effect on Cardiovascular Events (DECLARE)-TIMI 58 Diabetes Trial in Healthcare Claims
Brief Title: Replication of the DECLARE Diabetes Trial in Healthcare Claims
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-DECLARE
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dapagliflozin: Exposure group
  Interventions: Drug: Dapagliflozin
- DPP-4 inhibitor: Reference group
  Interventions: Drug: DPP-4 inhibitor

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin dispensing claim for any dose is exposure
  Groups: Dapagliflozin
Drug: DPP-4 inhibitor — DPP4 inhibitor dispensing claim for any dose is reference
  Groups: DPP-4 inhibitor

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates:

Market availability of dapagliflozin in the U.S. started on January 8, 2014.

* For Marketscan and Medicare: Jan 8, 2014-Dec 31, 2017 (end of data availability).
* For Optum: Jan 8, 2014-Mar 31, 2019 (end of data availability).

Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures (including run-in)
2. Female or male aged ≥ 40 years
3. Diagnosed with T2DM
4. High Risk for CV event defined as having either established CV disease and/or multiple risk factors:

   - Established CV Disease (See Appendix E for details) OR No known cardiovascular disease AND at least two cardiovascular risk factors in addition to

   T2DM, defined as:
   * Age > 55 years in men and > 60 in women AND presence of at least 1 of the following additional risk factors (see Appendix E for details)
   * Dyslipidemia
   * Hypertension
   * Tobacco use
5. WOCBP must take precautions to avoid pregnancy throughout the study and for 4 weeks after intake of the last dose.

   * WOCBP must have a negative urine pregnancy test. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal.
   * WOCBP must be willing to use a medically accepted method of contraception that is considered reliable in the judgment of the Investigator. For inclusion in the optional genetic research, patients must fulfill the criterion specified in

Exclusion Criteria:

Patients should not meet any exclusion criteria at the time of randomization. If at the time of enrollment, it is known that the patient will not meet criteria after a successful run-in period he/she should not be entered into run in.

1. Use of the following excluded medications:

   * Current or recent (within 24 months) treatment with pioglitazone and/or use of pioglitazone for 2 years or more at any time
   * Current or recent (within 12 months) treatment with rosiglitazone
   * Previous treatment with any SGLT2 inhibitor
   * Any patient currently receiving chronic (>30 consecutive days) treatment with an oral steroid at a dose equivalent to oral prednisolone ≥10 mg (e.g., betamethasone ≥1.2 mg, dexamethasone ≥1.5 mg, hydrocortisone ≥40 mg) per day
2. Acute cardiovascular event [e.g., acute coronary syndrome (ACS), transient ischemic attack (TIA), stroke, any revascularization, decompensated HF, sustained tachycardia <8 weeks prior to randomization. Patients with acute cardiovascular events can be enrolled in the run-in period as long as randomization does not occur within 8 weeks of the event.
3. Systolic BP >180 or diastolic BP >100 mmHg at randomization
4. Diagnosis of Type 1 diabetes mellitus, MODY, or secondary diabetes mellitus
5. History of bladder cancer or history of radiation therapy to the lower abdomen or pelvis at any time
6. History of any other malignancy within 5 years (with the exception of successfully treated non-melanoma skin cancers)
7. Chronic cystitis and/or recurrent urinary tract infections (3 or more in the last year)
8. Any conditions that, in the opinion of the Investigator, may render the patient unable to complete the study including but not limited to cardiovascular (NYHA class IV CHF, recurrent ventricular arrhythmias) or non-cardiovascular disease (e.g., active malignancy with the exception of basal cell carcinoma, cirrhosis, chronic lung disease, severe autoimmune disease) and/or a likely fatal outcome within 5 years
9. Pregnant or breast-feeding patients
10. Involvement in the planning and/or conduct of the study or other dapagliflozin studies (applies to AZ, BMS, Hadassah and Thrombolysis in Myocardial Infarction [TIMI] or representative staff and/or staff at the study site)
11. Previous randomization in the present study
12. Active participation in another clinical study with IP and/or investigational device
13. Individuals at risk for poor protocol or medication compliance during run-in period (reasonable compliance defined as 80 - 120%, unless a reason for non-compliance is judged acceptable by the Investigator). If for any reason, the Investigator believes that the patient will not tolerate or be compliant with IP or study procedures, the patient should not be randomized and considered a run-in failure. Patients will be excluded during run-in and should not be randomized if the following are observed from laboratory or observation during enrollment and run-in assessments:
14. HbA1c ≥12% or HbA1c<6.5%
15. AST or ALT >3x ULN or Total bilirubin >2.5 x ULN
16. CrCl < 60 ml/min (based on the Cockroft-Gault equation)
17. Hematuria (confirmed by microscopy at Visit 1) with no explanation as judged by the Investigator up to randomization. If bladder cancer is identified, patients are not eligible to participate.
18. Any reason the Investigator believes the patient is not likely to be compliant with the study medication and protocol.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing dapagliflozin to the DPP-4 inhibitor (DPP4i) antidiabetic class. DPP4is serve as a proxy for placebo, since this class of antidiabetic drugs is not known to have an impact on the outcome of interest. The comparison against DPP4 inhibitors is the primary comparison. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of canagliflozin or a comparator drug (cohort entry date). Follow-up for the outcomes (a. 3P-MACE and b. composite of heart failure hospitalization/all-cause mortality), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during the study.
Sampling Method: Non-Probability Sample
Enrollment: 49790 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Composite outcome of Stroke, MI, and Mortality | Through study completion (a median of 120-140 days)
  Composite outcome of MI, stroke, and mortality - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Womens
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Franklin JM, Patorno E, Desai RJ, Glynn RJ, Martin D, Quinto K, Pawar A, Bessette LG, Lee H, Garry EM, Gautam N, Schneeweiss S. Emulating Randomized Clinical Trials With Nonrandomized Real-World Evidence Studies: First Results From the RCT DUPLICATE Initiative. Circulation. 2021 Mar 9;143(10):1002-1013. doi: 10.1161/CIRCULATIONAHA.120.051718. Epub 2020 Dec 17. PMID 33327727

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT04215523/Prot_SAP_001.pdf